CLINICAL TRIAL: NCT01557478
Title: Melatonin in Improving the Quality of Life of Breast Cancer Patients and Reduction of Postoperative Pain and Chemotherapy Induced Toxicity
Brief Title: Melatonin as Adjuvant Therapy in Breast Cancer Patients
Acronym: MIQOL-B
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Khon Kaen University (Other)
Collaborators: National Research Council of Thailand (Other Government); Srinagarind Hospital, Khon Kaen University (Other); Maharat Hospital, Nakhon Ratchasima (Unknown); General Drugs House Co.,LTD. (Other)
Responsible Party: Principal Investigator, Nutjaree Pratheepawanit Johns, Associate Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIQOL-B
Record Dates: First submitted 2012-03-13; First posted 2012-03-19 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Stage II and III Breast Cancer
Keywords: breast cancer; melatonin; adjuvant therapy; quality of life; pain; sleep; survival; adverse events
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Matched placebo (Placebo Comparator): Matched placebo (identical formulation and delivery, without active ingredient)
  Interventions: Drug: match placebo
- Melatonin 20mg (Active Comparator): 20 mg melatonin gelatin capsule
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — 20 mg melatonin gelatin capsule (1) taken orally after 21:00 hours each night throughout the study
  Arms: Melatonin 20mg
Drug: match placebo — placebo gelatin capsule (1) taken orally after 21:00 hours each night throughout the study
  Arms: Matched placebo

SUMMARY:
The study evaluate the effect of melatonin in improving quality of life and reducing post operative pain and chemotherapy-induced toxicity in breast cancer patients. This is a multi-center, randomized, double-blind, placebo controlled trial conducted in stage II or III breast cancer patients. Mixed-block randomization, stratified by center and treatment scheme is used to divide eligible patients into two groups: melatonin 20 mg or matched placebo. The patients are required to take the studied drugs at night (after 21.00 pm) on the first night prior to surgery and continue for 24 months. Standard treatment is surgery followed by chemotherapy according to each center's standard protocol. Study endpoints are QOL (FACT-B), pain (VAS 0-10), adverse event frequency, sleep quality (VAS 0-10), recurrence rate and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven stage II or III breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
* platelet count ≥100,000 cells/mm3
* white blood cell count ≥ 3,000 cell/mm3
* hemoglobin ≥ 10 g/dL
* serum creatinine ≤ 1.5 mg/dL
* bilirubin ≤ 2 mg/dL
* AST ≤ 2.5 times upper limit of normal (ULN)
* New York Heart Association grade ≤ 2
* written consent

Exclusion Criteria:

* received prior chemotherapy or biotherapy, radiotherapy or surgery within 1 month preceding randomization,
* had more than one type of cancer or brain metastasis
* moderate neuropathy (CTCAE grade ≥ 2)
* active infection
* uncontrolled complications (i.e. blood glucose > 200 mg/dL, uncontrolled hypertension, unstable angina, history of congestive heart failure or history of myocardial infarction within one year).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-03; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (FACT-B Version 4) | Change from baseline in TOI scores at 6 months
  Self-reported questionnaire. FACT-B Thai Version 4 has been previously validated. Change from baseline will be evaluated at months 2,4,6,12,18,24.

SECONDARY OUTCOMES:
Pain and amount of pain medication used | Before and up to 72 hours after surgery.
  Self-reported VAS scale (0-10)
Number of participants with adverse events | Baseline and months 2,3,4,5,6,12,18,24
  CTCAE Version 4.3
Sleep quality | Baseline, up to 72 hours after surgery and months 2,3,4,5,6,12,18,24
  Self reported VAS scale (0-10)
Cancer recurrence incidence | participant will be followed for the duration of study, an expected average of 2 years
Progression-free survival | participant will be followed for the duration of study, an expected average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nutjaree P Johns, PharmD,PhD, Principal Investigator — Khon Kaen University
Locations (2):
- Thailand (2):
  - Srinagarind Hospital, Khon Kaen, Changwat Khon Kaen
  - Maharat Nakorn Ratchasima Hospital, Nakorn Ratchasima, Nakorn Ratchasima